CLINICAL TRIAL: NCT07167927
Title: Developing an Innovative Decision Support Tool for Pediatric Neuromuscular Scoliosis - Aims 2 and 3
Brief Title: Developing an Innovative Decision Support Tool for Pediatric Neuromuscular Scoliosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Jody Lin, MD, University of Utah
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB_00169930; 1K23AR079778 (NIH)
Record Dates: First submitted 2025-08-26; First posted 2025-09-11 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Children With Medical Complexity (CMC); Multiple Chronic Conditions; Neuromuscular Scoliosis; Shared Decision Making; Decision Support Systems, Clinical; Decision Aids
Keywords: children with medical complexity; shared decision making; values clarification; uncertainty communication; decision support tool
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Intervention Model Description: pre-intervention crossed over to post-intervention design for provider participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Participants receive usual care
- Decision support tool (Experimental): Participants receive the novel decision support tool
  Interventions: Behavioral: Decision support tool

INTERVENTIONS:
Behavioral: Decision support tool — Decision support tool developed for patients, parents, and providers of children with neuromuscular scoliosis
  Arms: Decision support tool

SUMMARY:
The goal of this pilot hybrid type I efficacy/implementation trial is to assess a newly developed decision support tool patients, parents, and providers to use during surgical treatment decision making for neuromuscular scoliosis (NMS). Results from this pilot will inform the design of a future larger effectiveness trial of the decision support tool.

Participants will either receive usual care or receive the decision support tool. Researchers will assess the decision made, decision quality, individual affective, cognitive, and behavioral effects, and feasibility and acceptability of tool use. They will also collect potential barriers and facilitators to implementation and feedback about the tool and study design to maximize likelihood of successful deployment of the tool into clinical practice and inform the design of a future trial. The outcomes measures will be used to inform potential effect size estimates to inform a future trial.

DETAILED DESCRIPTION:
Neuromuscular scoliosis (NMS) can result in severe disability for children. Non-operative management including bracing and physical therapy minimally slows scoliosis progression, but operative management with posterior spinal fusion (PSF) carries high risks of morbidity and mortality in part due to the multiple comorbid conditions seen in children with NMS. Decisions like PSF that have no clear best treatment option are best served by shared decision making (SDM). SDM is a collaborative process where patients, parents, and providers share their knowledge, preferences, and values to reach treatment plan agreement. Our prior qualitative study creating a framework of SDM for children with multiple comorbid conditions like children with NMS found that parents face immense decision related uncertainty that often goes unacknowledged by providers and that parents and providers struggle with identifying and communicating family preferences and values that are important for treatment decision making. Our prior work has identified optimal methods to communicate uncertainty and identified the preferences and values parents of children with NMS have when it comes to treatment decision making for NMS. This study will pilot test a decision support tool that contains these elements.

ELIGIBILITY:
Inclusion criteria:

* Parent-child dyads of children with neuromuscular scoliosis who speak English and Spanish.
* Child is between ages 8-21 years of age and they are coming into the pediatric orthopaedic surgery clinic for consultation about potential surgery for NMS.
* NMS is defined as having neurologic impairment (NI) and scoliosis using relevant ICD-9 or ICD-10 codes from Feudtner, et al. 2014 or Berry, et al. 2012. or a qualifying diagnosis per the Pediatric Spine Study Group definition of NMS.
* All pediatric orthopaedic surgeons and neurosurgeons who treat neuromuscular scoliosis at our study sites will be eligible participants.

Exclusion criteria:

* Families whose child with NMS is less than 8 years of age at time of orthopaedic consultation because surgery at a younger age usually indicates an atypical case.
* Children with the diagnosis of Duchenne's or Becker's muscular dystrophy due to potential disease modifying therapies that may alter curve progression.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Intention for NMS treatment | Immediately after clinic visit
  Parent degree of decision preference (1: no surgery-9: surgery)

SECONDARY OUTCOMES:
Intention for NMS treatment | Immediately after clinic visit
  Parent's desired treatment option: Binary (1- surgery, 0- no surgery)
Intention for not delaying treatment | Immediately after clinic visit
  For parents who select surgery, the intention of treatment timing.
Knowledge questions | Immediately after clinic visit
  Parent's response to five decision-related knowledge questions, scored as total answered correctly
Acceptability of intervention | Immediately after clinic visit
  Measured quantitatively by the validated Acceptability of Intervention Measure for caregivers in the intervention group. The scale consists of 4 items rated on a 5-point Likert scale. A mean score is created with a higher score indicating higher acceptability.
Physician trustworthiness | Immediately after clinic visit
  The Dugan Physician Trust Scale is a validated 5-item survey measure to assess the participant's trust in their physician. Each item is rated on a 5-point Likert scale and one item is reverse coded before all items are summed to create a composite score. Higher scores indicate stronger trust in the physician.
Feasibility of intervention | Immediately after clinic visit
  Measured by the validated Feasibility of Intervention Measure. The scale consists of 4 items rated on a 5-point Likert scale. A mean score is created with a higher score indicating higher acceptability.
Risk perception | Immediately after clinic visit
  2 unique items on perception of risk related to decision, scored individually. Each item is rated on a 5-point Likert scale. The items will be scored individually with higher responses indicating higher perceived decision-related risk.
Decision conflict | Immediately after clinic visit
  Decisional conflict scale and 2 unique decision conflict items (individual items scored individually). Each item is rated on a 5-point Likert scale. The items will be scored individually with higher responses indicating higher decisional conflict.
Decision readiness | Immediately after clinic visit
  Preparation for Decision Making (PrepDM):
  The PrepDM scale is a validated 10-item survey measure that evaluates the participant's perception of how helpful their clinic visit was in preparing them to make the decision. Each item is rated on a 5-point Likert scale, and scores are standardized to a 0-100 scale, with higher scores indicating greater perceived readiness for decision-making.
Acceptability of Intervention- Qualitative | Within 3 months of clinic visit (for parents) and at end of study, approximately within 18 months of consent (for providers).
  Qualitatively assessed via focus groups and individual interviews for caregivers in intervention group and provider participants.
Worry | Immediately after clinic visit
  Consists of 3 unique items to assess the participant's level of worry related to decision making. Each item is rated on a 5-point Likert scale. The items will be scored individually with higher responses indicating higher levels of decision-related worry.
Quality of shared decision making | Immediately after clinic visit
  Quantitatively via the 9-item SDM-Q-9 (parent) and SDM-Q-Doc (provider) surveys. Each item is rated on a 6-point Likert scale. The total score is standardized to a scale from 0 to 100, with higher scores indicating greater perceived involvement in decision-making.
Decisional self-efficacy | Immediately after clinic visit
  The Decisional Self-Efficacy Scale is a validated 11-item survey measure that evaluates the participant's ability to make informed health-related decisions. Items are rated on a 5-point Likert scale and scores are standardized to a 0-100 scale, with higher scores reflecting greater decisional self-efficacy.
preference concordance for parents | Immediately after clinic visit
  Compare parent self-rated top three values/preferences driving decision making with decision they chose for consistency of decision with values/preferences. Will be scored based on number of values (out of 3) that match the treatment option selected.
Appropriateness of intervention | Immediately after clinic visit
  Measured quantitatively by the validated Appropriateness of Intervention Measure. The scale consists of 4 items rated on a 5-point Likert scale. A mean score is created with a higher score indicating higher acceptability.
Preference concordance between parents and providers | Immediately after clinic visit
  Correlation between top three parent preferences and values for decision identified by parents and by providers, calculated via a kappa score.
Feasibility of Intervention- Qualitative | Within 3 months of clinic visit (for parents) and at end of study, approximately within 18 months of consent (for providers).
  Qualitatively assessed via focus groups and individual interviews for caregivers in intervention group and provider participants.
Appropriateness of Intervention- Qualitative | Within 3 months of clinic visit (for parents) and at end of study, approximately within 18 months of consent (for providers).
  Qualitatively assessed via focus groups and individual interviews for caregivers in intervention group and provider participants.
Quality of shared decision making- qualitative | During clinic visit
  Using the DEEP-SDM coding scheme on video- and audio-recorded clinical encounters

OTHER OUTCOMES:
Barriers and facilitators to implementation | Within 3 months of clinic visit (for parents) and at end of study, approximately within 18 months of consent (for providers).
  Qualitative analysis of interviews and focus groups from intervention group participants using the CFIR
Quality of interpretation | immediately after clinic visit
  5-item survey questions based on Napoles 2015 and qualitative analysis of recorded clinic visits to assess quality of interpretation. The first item assesses the type and need for interpretation, with participants selecting from 7 categories. If an interpreter was used, participants will then answer 4 additional items about the quality of interpretation for the visit. Each of these subsequent items is rated on a 5-point Likert scale (1-poor to 5-excellent). A mean composite outcome of the completed items is used to calculate overall quality.
Usability of intervention | Immediately after clinic visit
  System Usability Scale (SUS):
  The SUS is a validated 10-item survey measure that evaluates the perceived usability of the intervention. Items are rated on a 5-point Likert scale and scores are calculated by converting responses to a 0-100 scale, with higher scores indicating better usability. Only parent participants assigned to the intervention group will answer this measure.
Mental load of intervention | Immediately after clinic visit
  NASA Task Load Index (NASA-TLX):
  The NASA-TLX is a validated measure used to assess the perceived mental workload of using the intervention. It consists of 6-items to measure 6 core dimensions: mental demand, physical demand, temporal demand, performance, effort, and frustration. Each dimension is rated on a scale from 0 to 100, and scores are combined to produce an overall workload score. Higher scores indicate greater perceived workload. Only parent participants assigned to the intervention group will answer this measure.
Tool use | End of study, approximately 18 months after first enrollment.
  Metadata on tool interaction, inputs, and use
Severe pneumonia | Within 18 months of clinic visit
  Chart review of medical records to count number of admissions for pneumonia.
Readability | Immediately after the clinic visit
  Consists of 2 unique items to assess how clearly the intervention is presented. Each item is rated on a 5-point Likert scale. The items will be scored individually. Only parent participants assigned to the intervention group will answer these items.
provider preferences and values for decision making | immediately after clinic visit
  provider free response of top three reasons for decisiion that was made
parent preferences and values | immediately after visit
  selection of top three parent preferences and values for decision making from a list of options including a free response "other" field; asked to parent/patient participants and provider participants
Quality of interpretation | During clinic visit
  Qualitative analysis of quality of interpretation captured on video-recordings of clinic visits.
Decision adherence | Within 18 months after clinic visit.
  Chart review of medical records to assess adherence to decision made.
Pain symptoms | Within 18 months of clinic visit
  Chart review of patient record for changes in pain symptoms related to scoliosis. Options include: worsened, unchanged, improved, not mentioned.
Surgical outcomes | Within 18 months of clinic visit
  Chart review of medical records to assess for presence surgical outcomes: minor complications, major complications.
Sitting comfort | Within 18 months of clinic visit
  Chart review of patient record for changes in sitting comfort symptoms related to scoliosis. Options include: worsened, unchanged, improved, not mentioned.
ICU length of stay | Within 18 months of clinic visit
  For those who undergo surgery, the days the patient spent in the ICU after surgery
Total length of stay | Within 18 months of clinic visit
  For those who undergo surgery, the days the patient spent in the the hospital after surgery
Length of ventilation | Within 18 months of clinic visit
  For those who undergo surgery, the days the patient spent on mechanical ventilation (if not ventilated at baseline) or days spent on higher than normal mechanical ventilation settings (if ventilated at baseline).
Pneumonia hospital days | Within 18 months of clinic visit
  Chart review of medical records to count number of days admitted for pneumonia.

CONTACTS AND LOCATIONS:
Overall Officials: Jody Lin, MD, MS, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No